CLINICAL TRIAL: NCT05285462
Title: Feasibility of Virtual Reality Delivery of Pain Neuroscience Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Belmont University (Other); Benchmark Physical Therapy (Unknown)
Responsible Party: Principal Investigator, Elizabeth Lane, Co-Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00145358
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care PT (Active Comparator): Patients will attend normal course of PT without influence from study team.
  Interventions: Behavioral: Usual Care Physical Therapy
- Usual Care PT + VR Pain Education (Experimental): Patients will attend normal course of PT without influence of duration or frequency of care. Patients will also receive up to 12 session of pain education delivered via VR headset
  Interventions: Behavioral: VR Pain Education; Behavioral: Usual Care Physical Therapy

INTERVENTIONS:
Behavioral: VR Pain Education — pain education delivered via VR headset, up to 12 sessions
  Arms: Usual Care PT + VR Pain Education
Behavioral: Usual Care Physical Therapy — Normal course of PT without influence by study team on frequency or duration

SUMMARY:
Randomized Clinical Trail (RCT) for patients already planned to attend physical therapy for chronic low back pain. Patients will be randomized to receive Physical Therapy (PT) as usual or PT plus pain education delivered via virtual-reality headset.

DETAILED DESCRIPTION:
There is an increasing emphasis in physical therapy and healthcare in general on enhancing patients' ability to self-manage spinal pain as a strategy to reduce disability for impacted individuals and escalating healthcare costs. This change in emphasis requires a paradigm shift on the part of practitioners and patients alike in how they conceptualize and respond to pain. PNE is a promising education strategy that has been shown to influence patient-reported outcomes in those with chronic pain and has been shown to influence the provider's beliefs about pain. However, the delivery of this education has proven difficult for providers in terms of comfortability and time-efficiency. A standardized delivery a PNE by experts in the field could prove efficient and effective.

STUDY DESIGN The investigators' overall goal is to determine the feasibility of VR-delivered pain neuroscience education (PNE). Secondarily, the investigators would like to see if these interventions are best targeted to specific individuals. To accomplish these goals, the investigators will conduct a randomized clinical trial, randomly assigning participants to receive virtual reality (VR) education in addition to usual care or usual care with no additional education.

ELIGIBILITY:
Inclusion Criteria:

* i. Age 18-75 at time of first physical therapy session ii. Primary reason for physical therapy is low back pain iii. History of low back pain >/= 12 weeks

Exclusion Criteria:

* i. Age >75y/o or <18 y/o ii. Red flag condition that prohibits participation in physical therapy:

  * Systemic metabolic disorder
  * Neurological or muscular degenerative disorder (including Epilepsy)
  * Systemic infection
  * Cardiopulmonary or pulmonary disorder with contraindication to physical exercise iii. Recent spinal surgery (<12 months) iv. Specific spinal pathologies, such as severe stenosis or spondylolisthesis or fracture v. Acute radiculopathy or compromised nerve root vi. Currently known to be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Rate of Recruitment | 6 weeks
  Count of all potentially eligible subjects (count kept by office coordinators of patients offered the study); count of those determined eligible by research team; count of those that choose to consent. Reasons for no contact or choosing not to enroll will be collected when able.
Adherence | 6 weeks
  Number of visits completed, number of VR modules completed.
Acceptability Measures | 6 weeks
  Patient satisfaction and acceptability of VR-delivered PNE.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI | 6 weeks
  Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. The ODI shows good internal consistency (α=0.85). Discrimination of all the items is high to perfect (1.08-2.01).
Numeric Pain Rating Scale (NPRS) | 6 weeks
  ranges from 0 (no pain) to 10 (worst imaginable pain) as a measure of pain intensity. The NPRS has excellent test retest reliability for LBP (0.61) and neck pain (0.76).
Pain Self-Efficacy Questionnaire (PSEQ): | 6 weeks
  quantifies an individual's confidence in performing activities despite pain. The PSEQ contains 10 items ranked from 0 ("not at all confident") to 7 ("completely confident"). The PSEQ has high validity when compared with measures of coping (r=0.48) and pain beliefs (r=0.74) and excellent test-retest reliability (0.73).
Pain Catastrophizing Scale (PCS) | 6 weeks
  is used to quantify the catastrophic thoughts regarding pain. Scores range from 0 to 52, with higher scores indicating higher levels of pain catastrophizing. The PCS was found to be highly reliable (chronbach alpha=0.75 to 0.86) and have good criterion-related, concurrent, and discriminant validity.
Global Rating of Change (GROC | 6 weeks
  is used to gain the patient's perceived progress of their condition since the beginning of physical therapy. The GROC ranges from +7 (a very great deal better to 0 (about the same) to) -7(a great deal worse). The GROC is a valid measure of measuring a patient's perceived change in quality of life.
Neurophysiology of Pain Questionnaire (NPQ) | 6 weeks
  is used to gain information regarding the how the patient conceptualizes the origins of his/her pain. This this tool to has acceptable internal consistency and test-retest reliability.
Fear Avoidance Beliefs Questionnaire (FABQ) | 6 weeks
  is used to assess fear and avoidance beliefs related to physical activity (FABQ-PA) and work activity (FABQ-W).
Brief Resiliency Scale (BRS): | 6 weeks
  a measure of a person's ability to bounce back or recover from stress.
Back Beliefs Questionnaire (BBQ): | 6 weeks
  measure patient's attitudes and beliefs towards recovery and return-to-work; and expectations regarding the negative circumstances that could be created as a result of low back pain (LBP)
Working Alliance Inventory (WAI): | 6 weeks
  measure of the therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. We will be using the short-form version. (Hatcher 2006)

CONTACTS AND LOCATIONS:
Locations (1):
- Belmont University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No